CLINICAL TRIAL: NCT01903525
Title: Docosahexaenoic Acid (DHA) For The Treatment of Pediatric Concussion Related to Sports Injury
Brief Title: DHA For The Treatment of Pediatric Concussion Related to Sports Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other); Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Principal Investigator, Shane M. Miller, MD, MD, Associate Professor of Orthopaedics and Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 042012-055
Record Dates: First submitted 2013-07-09; First posted 2013-07-19 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Concussion; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo capsules are supplied as 950 mg capsules consisting of 475 mg corn oil and 475 mg soy oil. Both DHA and placebo are flavored with sweet orange flavoring and masking agents. Subjects will be instructed to take 2 capsules at breakfast and 2 capsules at dinner (with food). Subjects will take their first dose in the office to assure their ability to swallow the pills. Subjects will be dosed with the placebo for 12 weeks.
  Interventions: Drug: Placebo
- Docosahexaenoic Acid (DHA) (Experimental): The DHASCO capsules are supplied as 950 mg capsules with an effective dose of 500 mg DHA per capsule. Both DHA and placebo are flavored with sweet orange flavoring and masking agents. Subjects will be instructed to take 2 capsules at breakfast and 2 capsules at dinner (with food). Subjects will take their first dose in the office to assure their ability to swallow the pills. Subjects will be dosed with the DHA for 12 weeks.
  Interventions: Drug: Docosahexaenoic acid (DHA)

INTERVENTIONS:
Drug: Docosahexaenoic acid (DHA) — Subjects presenting with a new concussion within 4 days of their initial injury will be identified and screened for eligibility from the investigators' regularly scheduled clinic patients. Subjects who enroll will complete 5 scheduled visits, although additional visits may be clinically indicated for symptom evaluation and treatment. All assessments done for this study are routinely done as part of the standard clinic visits for concussion at the Sports Medicine Center. Subjects will be randomized to either DHA or placebo in a 1:1 ratio, and receive enough DHA or placebo capsules to reach the target dose of 2 g of DHA per day (or placebo) until the day of their next appointment. Subjects will be instructed to take 4 capsules (2 at breakfast and 2 at dinner) for 12 weeks.
  Arms: Docosahexaenoic Acid (DHA)
Drug: Placebo — Subjects presenting with a new concussion within 4 days of their initial injury will be identified and screened for eligibility from the investigators' regularly scheduled clinic patients. Subjects who enroll will complete 5 scheduled visits, although additional visits may be clinically indicated for symptom evaluation and treatment. All assessments done for this study are routinely done as part of the standard clinic visits for concussion at the Sports Medicine Center. Subjects will be randomized to either DHA or placebo in a 1:1 ratio, and receive enough DHA or placebo capsules to reach the target dose of 2 g of DHA per day (or placebo) until the day of their next appointment. Subjects will be instructed to take 4 capsules (2 at breakfast and 2 at dinner) for 12 weeks.
  Arms: Placebo

SUMMARY:
In recent years, media attention has focused on the long-term sequelae of repeated concussive episodes in professional athletes. The growing understanding of the damage done by what was once considered a "ding" during a game or match, and the neurologic consequences of "playing through" or returning to play too soon has led to additional interest in and concern for pediatric athletes (18 or under) who experience sports-related concussions during game or practice play.

Because it has only been in recent years that the full scope of damage done by repeated concussive episodes has come to light, very little research has been done on treatment of concussion in either adults or children. Brain injuries in children can be especially problematic, as the brain may continue to develop until the child reaches the age of 24 or older, so concussion during this time of development may be particularly damaging.

Docosahexaenoic acid (DHA) is an omega-3 fatty acid commonly found in both fish oils and algae. DHA is known to improve development of the eyes and brain in young children. It is thought to be an effective anti-inflammatory and anti-oxidant, and since it occurs naturally and causes very few harmful side effects, it may be a useful compound in the treatment of pediatric concussion.

This is a feasibility trial of DHA for the treatment of sports concussion in a pediatric population. The investigators' primary aim is to determine acceptability of randomization for this compound as well as rate of enrollment given our clinical population. The investigators' secondary aim is to examine preliminary outcomes. The investigators hypothesize that subjects who take 2 g of DHA daily for 3 months will see a shorter time to full recovery and return to play and a shorter time to resolve balance disturbance. These are good, albeit unvalidated, clinical indicators of concussive recovery.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled feasibility trial of DHA for the treatment of pediatric concussion related to sports-injury. The definition used for concussion is from the Consensus Statement on Concussion in Sport: the 3rd International Conference on Concussion in Sport (Br J Sports Med 2009;43:Suppl 1 i76-i84 doi:10.1136/bjsm.2009.058248) and will meet the following criteria:

1. Direct blow to the head, face, neck or a blow elsewhere on the body with an "impulsive" force transmitted to the head.
2. Rapid onset of short-lived impairment of neurologic function in one or more of the following clinical domains that resolves spontaneously:

   1. symptoms: somatic (eg, headache), cognitive (eg, feeling like in a fog) and/or emotional symptoms (eg, lability).
   2. physical signs (eg, loss of consciousness, amnesia).
   3. behavioural changes (eg, irritability).
   4. cognitive impairment (eg, slowed reaction times).
   5. sleep disturbance (eg, drowsiness).
3. No abnormality on standard structural neuroimaging studies, if such neuroimaging studies are completed for a clinically-indicated reason. Note: neuroimaging is not a part of this study protocol. Study participants will not undergo neuroimaging as part of this study.

Subjects will be randomized in a 1:1 fashion. DHA is an omega-3 fatty acid that occurs naturally in fish oil and algae. There are many dietary supplements containing DHA available in the marketplace. Martek Biosciences provides an algae-based DHA compound which minimizes the side effects of "fishiness" in both flavor and "fish burps." The DHA produced by Martek Biosciences is also used for many infant formula companies in the US. DHA and identical placebo will be provided by Martek Biosciences.

The DHASCO capsules are supplied as 950 mg capsules with an effective dose of 500 mg DHA per capsule. The placebo capsules are supplied as 950 mg capsules consisting of 475 mg corn oil and 475 mg soy oil. Both DHA and placebo are flavored with sweet orange flavoring and masking agents.

They are supplied in sealed white plastic bottles containing 100-200 capsules per bottle, depending on dose. Each bottle has the lot number stamped on it. The capsules will be stored in a dry, locked compartment at room temperature (60 to 75 F). Martek's Quality Assurance department completes regularly scheduled chemical and long-term stability analyses on each lot of capsules. If shipments will occur during warmer months, arrangements will be made for capsules to be shipped with ice packs or other temporary refrigeration. Capsules will be dispensed to subjects in separate bottles in quantities sufficient to last until their next appointment. Any unused capsules will be returned to the PI or research staff and sent to the pharmacy for destruction in compliance with Children's regulations.

Subjects will be randomized to 2 g of DHA or matched placebo for 12 weeks. In order to achieve this dose of DHA, subjects will receive 2 950 mg capsules twice a day. Subjects who cannot tolerate the divided dose of 2000 mg per day will be discontinued from the study.

Although much of our knowledge of the pathophysiology of concussion comes from animal models, it is believed that the mechanical trauma to the brain causes a sudden disruption in the ionic balances, leading to an increase in calcium and an increase in glucose metabolism as cells try to compensate for the potassium/calcium imbalance. This is followed by a period of decreased glucose metabolism which may last up to 4 weeks in humans, resulting in continued high levels of calcium which interfere with mitochondrial oxidative metabolism. This decrease in mitochondrial oxidative metabolism appears to be biphasic, with improvement seen at 2, followed by a decrease which bottoms out on day 5 and recovers around day 10. Other important aspects of the concussive trauma include free radical production, initiation of inflammatory responses, and altered neurotransmission.

DHA has several important functions in the brain with relatively few side effects, making it a good option for concussion treatment. DHA is helpful in modulating ion channels; higher levels of DHA are associated with higher levels of sodium pump activity, so it is possible that providing DHA post-injury may help the cells reduce the calcium balance more quickly or efficiently. DHA also has an apparent anti-inflammatory action. DHA interferes with the inflammatory arachidonic acid cascade by reducing the affinity of platelet thromboxane A2/prostaglandin H2 (TxA2/PGH2) receptor for its ligand. Additionally, higher levels of DHA in the cerebral cortex cause significantly higher levels of the anti-oxidant enzymes catalase, glutathione and glutathione peroxidase -- resulting in decreased cerebral levels of lipid peroxides. DHA reduces formation of the peroxynitrite free radical and reduces formation of pro-inflammatory cytokines by inhibiting transcription factor NF-κB and inducible nitric oxide synthetase. Finally, DHA is highly concentrated in synapses, indicating a role in synaptic signal transduction. DHA appears to address many different aspects of how we believe concussive injury affects the brain.

The primary outcomes of this feasibility trial are to determine the willingness of patients to be randomized, the expected rate of enrollment based on the clinic population, and protocol adherence of enrolled study participants. We anticipate the results from this study will provide data to inform a larger randomized trial of DHA for the treatment of pediatric sports concussion. Secondary outcomes are time to clearance to return to play (in days) and improvement in balance, as assessed by the Balance Error Scoring System (BESS) which is a component of the Sport Concussion Assessment Tool 3 (SCAT-3). Time to clearance to return to play was chosen as a clinically significant measurement for medical professionals in the sports medicine field. The investigators will determine clearance for return to full competitive game play (Stage 6 of graduated return to play protocol) according to Consensus Statement guidelines and following the law in Texas, House Bill 2038. Criteria for return to play include complete clinical recovery from the concussion including returning to baseline symptoms, exam and neurocognitive function and successful completion of a gradual return to play progression. The BESS was chosen because it is a relatively simple assessment that has been noted by the investigators to be a good predictor of neurological recovery.

In addition to time to return to play and the BESS, the SCAT-3 and Immediate Post Concussion Assessment and Cognitive Testing (ImPACT) computerized neurocognitive testing programs will be used to evaluate recovery. The SCAT-3 is a standardized method of evaluating injured athletes for concussion and can be used in athletes aged from 10 years and older. The ImPACT program is a computerized exam that helps to quantify the degree of symptom, injury, or dysfunction that occurs after a sports related concussion. Although this test is utilized by many professionals, college, and high school sports programs throughout the country, it is unclear if its use contributes to a safer or more expedited return to activity.

Finally, information on side effects will be collected at every visit in order to track the rate and severity of side effects in this patient population.

We plan to enroll 40 subjects for this study, which consists of 20 subjects to be treated with DHA and 20 subjects to be treated with placebo. In order to achieve enrollment of 40 total subjects, we anticipate screening 80 subjects in order to consent 40. Because this is a pilot study, information on early withdrawals is important to us and no extra subjects will be consented due to this. We anticipate that it will take approximately 12 months to complete enrollment, with an additional 3 months for patient follow-up once the last patient has been enrolled. We anticipate that it will take approximately 6-9 months to complete data clean-up, analysis, and manuscript submission for total study duration of 2 years.

Subjects who are non-compliant with the protocol either by not keeping appointments or by not taking study pills as directed may be discontinued from the study. Subjects who do not tolerate the minimum dose of 2000 mg of DHA per day or who experience intolerable side effects will be discontinued. Subjects who choose to withdraw consent will be discontinued early.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females age 14-18 inclusive
2. Diagnosed with concussion due to sports-related injury. Concussion is defined as:

   1. Direct blow to the head, face, neck or a blow elsewhere on the body with an "impulsive" force transmitted to the head.
   2. Rapid onset of short-lived impairment of neurologic function in one or more of the following clinical domains that resolves spontaneously:

   i. Symptoms: somatic (eg, headache), cognitive (eg, feeling like in a fog and/or emotional symptoms (eg, lability).

   ii. Physical signs (eg, loss of consciousness, amnesia).

   iii. Behavioral changes (eg, irritability).

   iv. Cognitive impairment (eg, slowed reaction times).

   v. Sleep disturbance (eg, drowsiness). c) No abnormality on standard structural neuroimaging studies, if such neuroimaging studies are completed for a clinically-indicated reason. Note: neuroimaging is not a part of this study protocol. Study participants will not undergo neuroimaging as part of this study.
3. Concussion within 4 days of enrollment
4. Presenting for treatment to the Sports Medicine Center at Children's Medical Center

Exclusion Criteria:

1. Subjects not actively participating in an organized sport at time of enrollment
2. Subjects who received a concussion from an event other than playing a sport (motor vehicle accident, fall, etc.)
3. Subjects who participate in or received a concussion during participation in motorized sports (i.e., motorcross, dirt biking, jet skiing, etc.)
4. Subjects with radiographic evidence of traumatic brain injury (i.e., skull fracture, intracranial hemorrhage, cerebral contusion, etc).
5. Subjects with a prior diagnosed concussion in the previous 6 months.
6. Pregnant women.
7. Subjects sensitive to aspirin
8. Subjects diagnosed with high blood pressure and currently being treated with blood pressure medications
9. Subjects allergic to soy bean oil or corn oil.
10. Subjects currently taking fish oil or DHA supplements.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shane Miller, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Sports Medicine at Texas Scottish Rite Hospital for Children, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller SM, Zynda AJ, Sabatino MJ, Jo C, Ellis HB, Dimeff RJ. A Pilot Randomized Controlled Trial of Docosahexaenoic Acid for the Treatment of Sport-Related Concussion in Adolescents. Clin Pediatr (Phila). 2022 Nov;61(11):785-794. doi: 10.1177/00099228221101726. Epub 2022 Jun 19. PMID 35722886

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The placebo capsules are supplied as 950 mg capsules consisting of 475 mg corn oil and 475 mg soy oil. Both DHA and placebo are flavored with sweet orange flavoring and masking agents. Subjects will be instructed to take 2 capsules at breakfast and 2 capsules at dinner (with food). Subjects will take their first dose in the office to assure their ability to swallow the pills. Subjects will be dosed with the placebo for 12 weeks.
  Docosahexaenoic acid (DHA): Subjects presenting with a new concussion within 4 days of their initial injury will be identified and screened for eligibility from the investigators' regularly scheduled clinic patients. Subjects who enroll will complete 5 scheduled visits, although additional visits may be clinically indicated for symptom evaluation and treatment. All assessments done for this study are routinely done as part of the standard clinic visits for concussion at the Sports Medicine Center. Subjects will be randomized to either DHA or placebo in a 1:1 ratio, and receive enough DHA or placebo capsules to reach the target dose of 2 g of DHA per day (or placebo) until the day of their next appointment. Subjects will be instructed to take 4 capsules (2 at breakfast and 2 at dinner) for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Started | 20 | 20
Completed | 15 | 10
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 5 | 9
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Docosahexaenoic Acid (DHA) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.97 (1.03) | 16.02 (1.19) | 16.00 (1.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 15 | 14 | 29
  Race/Ethnicity: Unknown | 3 | 5 | 8
  Race/Ethnicity: Black or African American | 2 | 0 | 2
  Race/Ethnicity: Hispanic or Latino | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: One patient was missing height in their record, therefore, BMI could not be calculated.
  kg/m^2
    number analyzed (Participants) | 20 | 19 | 39
    (all) | 23.3 (3.2) | 25.0 (5.8) | 24.16 (4.74)
History of Previous Concussions [Count of Participants; unit: Participants]
  No | 11 | 17 | 28
  Yes | 9 | 3 | 12
Sport Injured [Count of Participants; unit: Participants]
  American Football | 8 | 9 | 17
  Soccer | 4 | 3 | 7
  Volleyball | 2 | 3 | 5
  Wrestling | 3 | 0 | 3
  Basketball | 0 | 2 | 2
  Softball | 1 | 1 | 2
  Lacrosse | 1 | 1 | 2
  Baseball | 1 | 0 | 1
  Karate | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of Higher Dosage of DHA
Description: Determine the safety of a higher dosage of DHA through reported drug-related adverse events during the study period.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 20 | 20
Participants | 0 | 1

2. Secondary Outcome: Drug Adherence During Study Period
Description: Determine the protocol treatment adherence/compliance of enrolled study participants.
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: percentage of adherence
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 20 | 20
percentage of adherence | 84.0 (9.1) | 74.7 (19.4)

3. Secondary Outcome: Time to Initiation of the Return to Sport (RTS) Progression
Description: Time to initiation of the return to sport progression (in days) was determined by calculating days from injury to when the participant was cleared to begin the return to sport progression by the physician. Time to initiation to return to sport progression was chosen as a clinically significant measurement for medical professionals in the sports medicine field. The investigators will determine time to initiation to return to sport progression according to Consensus Statement guidelines and following the law in Texas, House Bill 2038. Criteria for return to play progression include returning to baseline symptoms, exam and neurocognitive function. We hypothesize that participants who take 2g of DHA daily will experience no significant differences in recovery time when compared to participants who take a placebo.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 20 | 20
days | 19.5 [9 to 39] | 14.0 [8 to 66]

4. Secondary Outcome: Resolution of Balance Impairment
Description: Improvement in balance impairment associated with the injury, as assessed by the modified Balance Error Scoring System (mBESS) which is a component of the Sport Concussion Assessment Tool 3 (SCAT-3). We hypothesize a shorter time to resolve balance disturbance associated with the treatment of DHA. The mBESS is scored from 0-30 errors, with higher scores indicated a worse outcome (more errors).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 20 | 20
score on a scale
  Enrollment | 4.15 (2.46) | 4.45 (2.44)
  1-week Visit | 3.21 (2.42) | 3.5 (2.5)
  2-week Visit | 3.94 (2.93) | 2.7 (1.64)
  4-week Visit | 2.67 (2.12) | 1.75 (1.26)
  12-week Visit | 2.31 (1.55) | 2.57 (2.15)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each time point: enrollment, 1-week, 2-week, 4-week, 12-week follow-up visits.
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Docosahexaenoic Acid (DHA) (N=20)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT01903525/Prot_SAP_000.pdf